CLINICAL TRIAL: NCT07262554
Title: Evaluation of N-acetylcysteine as an Intracanal and Adjunctive Systemic Medication in Root Canal Treatment of Necrotic Mature Teeth With Apical Periodontitis: a Randomized Controlled Clinical Trial
Brief Title: N-acetylcysteine for Root Canal Treatment of Necrotic Teeth With Apical Periodontitis
Acronym: NAC
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, Mai Hussein, Assistant lecturer, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 9258326; PACTR202511513893768 (Registry Identifier: The Pan African Clinical Trial Registry (PACTR))
Record Dates: First submitted 2025-11-20; First posted 2025-12-03 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-11

CONDITIONS: Apical Periodontitis
Keywords: N-acetylcysteine (NAC); Calcium hydroxide (Ca(OH)₂); Intracanal medication; Root canal treatment; Apical periodontitis; Postoperative pain; Periapical healing; Periapical tissue biomarkers; Cone-beam computed tomography (CBCT)
MeSH Terms: conditions — Periapical Periodontitis; Pain, Postoperative | interventions — Calcium Hydroxide; Acetylcysteine

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two groups. Group I (control group): UltraCal XS calcium hydroxide (Ca(OH)₂) intracanal medication for 7 days; and Group II: N-acetylcysteine (NAC) intracanal medication for 7 days and 600 mg/day oral NAC for 21 days.
Who Masked: Outcomes Assessor
Masking Description: Two blinded and trained researchers, not involved in the intervention, will independently assess the pre- and postoperative radiographs. A blinded assessor will also perform the data analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Calcium hydroxide (Ca(OH)₂) (Active Comparator): UltraCal XS calcium hydroxide (Ca(OH)₂) intracanal medication for 7 days
  Interventions: Drug: Calcium hydroxide (Ca(OH)₂)
- N-acetylcysteine (NAC) (Experimental): N-acetylcysteine (NAC) intracanal medication for 7 days and 600 mg/day oral NAC for 21 days
  Interventions: Drug: N-Acetylcysteine (NAC)

INTERVENTIONS:
Drug: Calcium hydroxide (Ca(OH)₂) — UltraCal XS calcium hydroxide (Ca(OH)₂) intracanal medication for 7 days
  Arms: Calcium hydroxide (Ca(OH)₂)
Drug: N-Acetylcysteine (NAC) — N-acetylcysteine (NAC) intracanal medication for 7 days and 600 mg/day oral NAC for 21 days
  Other Names: Acetylcysteine; N-Acetyl-L-cysteine
  Arms: N-acetylcysteine (NAC)

SUMMARY:
A randomized controlled trial comparing the postoperative pain intensity, periapical biomarkers level, and periapical healing in patients with necrotic mature teeth and apical periodontitis treated with N-acetylcysteine (NAC), as an intracanal and adjunctive systemic medication, versus calcium hydroxide (Ca(OH)₂) intracanal medication alone.

ELIGIBILITY:
Inclusion Criteria:

* Mature necrotic teeth.
* Radiographic evidence of periapical bone loss.
* Teeth that require primary endodontic treatment.
* Restorable teeth.

Exclusion Criteria:

* Immature teeth
* Teeth that had been previously accessed or endodontically treated.
* Teeth with periodontal pockets deeper than 4 mm.
* Patients with acute apical abscess.
* Patients with systemic diseases.
* Pregnant females.
* Patients who received antibiotic therapy within the past month.
* Patient on analgesics.

Ages: 16 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2025-11-15 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Postoperative pain intensity | Pain will be recorded before the intervention, and patients will use the Numerical Rating Scale (NRS) to self-assess postoperative pain at 6 hours, 12 hours, 24 hours, 48 hours, 72 hours, and 1 week.
  Postoperative pain will be assessed using the Numerical Rating Scale (NRS), which is a scale from 0 (no pain) to 10 (worst pain imaginable). Patients will be asked to choose the number that represents their pain intensity. Pain level will be assigned as follows: 0, "no pain"; 1-3, "mild pain"; 4-6, "moderate pain"; 7-10, "severe pain."
Assessment of periapical healing | A CBCT scan will be taken preoperatively and at six months follow-up.
  Assessment of the percentage change in lesion volume through three-dimensional (3D) reconstruction of the lesions in Cone beam computed tomographic (CBCT) scans performed preoperatively and after a six-month follow-up.

SECONDARY OUTCOMES:
Change in the level of periapical tissues biomarkers | Samples will be collected from the periapical tissue fluid at two different points: before (S1) and after 7 days of administration of medications (S2).
  The biomarker levels will be measured using enzyme-linked immunosorbent assay [ELISA]. Samples of periapical tissue fluid will be taken by inserting three sterile paper points into the root canal, about 2 mm beyond the working length, and holding them in place for 1 minute. The paper points will be transferred to a 1.5-mL Eppendorf and stored at -80°C until further analysis.

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Alexandria University, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No